CLINICAL TRIAL: NCT06662565
Title: Effect of Pelvic Floor Down-training on Women With Idiopathic Overactive Bladder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ayatullah Farouk Abdelfattah Ahmed, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005319
Record Dates: First submitted 2024-10-26; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral modification group (Active Comparator): They will be treated with behavioral modification for 8 weeks.
  Interventions: Behavioral: Behavioral modification
- Pelvic floor down training and behavioral modification group (Experimental): They will be treated with the same behavioral modification plus pelvic floor down training three times per week for 24 sessions for 8 weeks.
  Interventions: Behavioral: Behavioral modification; Other: Pelvic floor down-training

INTERVENTIONS:
Behavioral: Behavioral modification — It includes:
  .- Reducing or eliminating smoking and carbonated drinks.
  * Weight loss in overweight or obese individuals.
  * Caffeine Reduction: Limiting caffeine intake, especially for those consuming at least 400 mg per day.
  * Consume Adequate Water: 6 to 8 glasses of water per day.
  * Refrain from consuming fluids 2 to 3 hours before bedtime.
  * Identify Bladder Irritants: such as sugar substitutes, citrus fruits, and tomato.
  * Increasing fiber intake like fruits, and vegetables to reduce constipation with adequate hydration to make stools softer and easier to pass
Other: Pelvic floor down-training — Pelvic floor down training exercises aimed at promoting relaxation and deconditioning of the pelvic floor muscles (PFM). It will be practiced three sessions per week for 8 weeks.
  Biofeedback-Assisted pelvic floor down-training:
  Procedure:
  * Rectal biofeedback will be inserted.
  * The therapist asks the woman to focus on consciously relaxing and releasing the PFM after each contraction or exercise while watching biofeedback screen.
  * Then, breathe deeply and fully into her abdomen, allowing her pelvic floor to naturally relax and lengthen.
  * And to incorporate relaxation techniques such as visualization, or progressive muscle relaxation to promote overall muscle relaxation and reduce PFM tension.
  * Exercises are typically repeated around 10-20 times per session. This number can vary depending on the patient's condition and tolerance, as well as the therapist's assessment and treatment plan.
  Arms: Pelvic floor down training and behavioral modification group

SUMMARY:
This study will be conducted to investigate the effect of pelvic floor down-training on women with idiopathic overactive bladder

DETAILED DESCRIPTION:
The relationship between overactive bladder (OAB), constipation, and overactive pelvic floor muscles is complex and interrelated. OAB increases the likelihood of overactive pelvic floor muscles, and conversely, hyperactive pelvic floor muscles can exacerbate OAB symptoms. Non-relaxing pelvic floor dysfunction often presents with urinary symptoms, including increased frequency, hesitancy, urgency, dysuria, bladder pain, and occasionally urge incontinence Pelvic floor down-training exercises targeting the rectum provide a safe, conservative way to manage constipation, which may in turn help relieve OAB. Unlike medications or surgery; these exercises are generally safe and easy to incorporate into daily life. However, more studies are needed to evaluate their effectiveness, especially for treating idiopathic OAB in women. Filling this research gap will provide clearer clinical guidance on managing the interplay between OAB, constipation, and pelvic floor hyperactivity. So this study will be the first to investigate the effect of pelvic floor down-training on symptoms of idiopathic OAB in women.

ELIGIBILITY:
Inclusion Criteria:

* Multiparous woman with idiopathic OAB (2-3 times) who diagnosed by physician and confirmed by the urodynamic study.
* Woman with high rectal resting tone measured by pressure biofeedback.
* Woman diagnosed with constipation according to the Rome IV criteria and Bristol score.
* Ages ranging from 30 to 45 years.
* BMI from 25-29.9 Kg/m2

Exclusion Criteria:

Women will be excluded from the study if they have:

* Severe OAB as measured by the overactive bladder symptom score for severity
* Postmenopausal women (a point in time 12 months after a woman's last period.)
* Any abnormalities around the bladder, such as bladder cancer, bladder calculus, interstitial cystitis, or endometriosis.
* Untreated urinary tract infections.
* Psychological or mental health problems.
* Pregnancy and lactation
* A history of previous pelvic surgery.
* Are receiving any pharmacological treatment at the time of the study.

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2024-10-31 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Rectal resting pressure | 8 weeks
  Biofeedback with intra-rectal probe (Myo200 manometer produced by Gymna. Bilzen. Belgium) will be used to measure rectal resting pressure before and after treatment for all women in both groups. Resting pressure is a good reflection of internal anal sphincter tone. The high resting pressure measures indicate pelvic floor hypertonicity which can indicate the presence of constipation.
Rectal bearing pressure | 8 weeks
  Biofeedback with intra-rectal probe (Myo200 manometer produced by Gymna. Bilzen. Belgium) will be used to measure rectal pressure during the bear-down maneuver before and after treatment for all women in both groups. the high pressure is an indicative of obstructed defecation.
Overactive Bladder Symptom Score (OABSS): | 8 weeks
  It will be used for assessing the severity of bladder symptoms before and after treatment for all women in both groups. The OABSS is validated, correlates well with other measures, and has high reliability. it measures the severity of overactive bladder symptoms like daytime frequency, nocturia, urgency, and urge incontinence. After the patient finishes the questionnaire, it will be collected for scoring, with each symptom scored separately and a total score calculated. The general score will be classified into three severity categories based on the total score: mild (0-5), moderate (6-11), and severe (12-20).
Assessment of overactive bladder symptoms | 8 weeks
  The Overactive Bladder Assessment Tool (OAB-BAT) evaluates bladder symptoms before and after treatment for all women in both groups. The OAB-BAT demonstrates strong construct validity and high reliability. It assesses frequency, urgency, and incontinence. It consists of 5 questions ranging from 0 to 5 for each. the higher scores indicating more severe symptoms.
Assessment of quality of life | 8 weeks
  The Overactive Bladder Assessment Tool (OAB-BAT) evaluates the quality of life of women with overactive bladder before and after treatment in both groups. The OAB-BAT demonstrates strong construct validity and high reliability. It consists of 6 questions ranging from 0 to 5 for each. the higher scores indicate poor quality of life.
Constipation scoring system | 8 weeks
  It is a questionnaire designed to evaluate the severity of constipation and has the advantage of not requiring digital rectal examination. It is valid and reliable and has a score ranging from 0 (minimum) and 30 (maximum), the higher the score, the more the severity of constipation symptoms.
Five-item score for obstructed defecation syndrome (ODS-S) | 8 weeks
  The questionnaire consists of 5 items: excessive straining, incomplete rectal evacuation, use of enemas and/or laxatives, vaginal-anal-perineal digitations, and abdominal discomfort and/or pain. Each item was graded from 0 to 5 with a score ranging from 0 (no symptoms) to 20 (very severe symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Amira N. Abdel Latif, PHD, Study Director — Cairo University; Doaa A. Osman, professor, Study Chair — Cairo University
Locations (1):
- Ayatullah Farouk Abdel Fattah, Cairo, Egypt